CLINICAL TRIAL: NCT01740986
Title: Double Blinded, Randomized, Placebo Controlled, Multi-center, Phase II Exploratory Clinical Study to Evaluate the Efficacy, Dose-response and Safety of SA09012 in Bronchial Asthma Patients
Brief Title: Safety and Efficacy of SA09012 in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SamA Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA09012-P2
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-01

CONDITIONS: Mild to Moderate Bronchial Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- SA09012 Low dose (Experimental)
  Interventions: Drug: SA09012 Low dose
- SA09012 High dose (Experimental)
  Interventions: Drug: SA09012 High dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SA09012 Low dose — Tablet, b.i.d
  Arms: SA09012 Low dose
Drug: SA09012 High dose — Tablet, b.i.d
  Arms: SA09012 High dose
Drug: Placebo — Tablet, b.i.d
  Arms: Placebo

SUMMARY:
Clinical Study to Evaluate the Efficacy, Dose-response and Safety of SA09012 in Bronchial Asthma Patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or presence of asthma within 3 months of the prestudy visit

  1. Increase in PEF ≥ 20% or ≥ 60L/min from baseline value after taking Bronchodilator at screening or within the 3 months of the prestudy visit
  2. Increase in FEV1 ≥ 12% and ≥ 200mL from baseline value after taking Bronchodilator at screening or within the 3 months of the prestudy visit
* FEV1 or PEF between 60% and 85% of the predicted value at screening or within the 3 months of the prestudy visit
* Having signed an informed consent

Exclusion Criteria:

* Patient who has severe asthma
* Patient who has any significant medical condition that might compromise patient safety, interfere with evaluation or preclude completion of the study other protocol-defined inclusion/exclusion criteria may apply
* Patient with an AST or ALT > 2x ULN (upper limit of normal) in the screening visit
* Patient with more than 10 pack year of cigarettes history

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline of PEF(Peak Expiratory Flow)at week 6 | 6 week treatment period

SECONDARY OUTCOMES:
Mean change from baseline in FEV1 at week 6 | 6 week treatment period
Mean change from baseline in ACT(Asthma Control Test) at week 6 | 6 week treatment period
Safety assessment(Comparison of the adverse event profiles throughout the course of the study) | 6 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Young Kyoon Kim, MD, Principal Investigator — Seoul ST. Mary's Hospital The Catholic University of Korea
Locations (14):
- South Korea (14):
  - Chonbuk National University Hospital, Chonbuk
  - Chonnam National University Hospital, Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - Bucheon St. Mary's Hospital, The Catholic University of Korea, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Gyeonggi-do
  - Chungbuk National University Hospital, Jungbuk
  - Konkuk University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Soonchunhyang University Hospital, Seoul, Seoul
  - St. Paul's Hospital, The Catholic University of Korea, Seoul
  - Yonsei University, Gangnam Severance Hospital, Seoul